CLINICAL TRIAL: NCT05253287
Title: Impact of Repurposed Growth Hormone Treatment on Clinical, Nutritional, Immunological and Regenerative Parameters in Decompensated Liver Cirrhosis: a Randomized Control Trial
Brief Title: Growth Hormone in Decompensated Liver Cirrhosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Nipun Verma, Assistant professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC-06/2021-2015
Record Dates: First submitted 2021-12-15; First posted 2022-02-23 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Liver Cirrhosis; Fibrosis; End Stage Liver Disease; Digestive System Disease; Physiological Effect of Drugs; Growth Hormone Treatment; Sarcopenia
Keywords: Decompensated liver cirrhosis; Growth hormone
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis; End Stage Liver Disease; Digestive System Diseases; Sarcopenia | interventions — Growth Hormone

STUDY DESIGN:
Intervention Model Description: Group 1 - Growth Hormone + Standard medical therapy Group 2 - Standard Medical Therapy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical treatment (No Intervention): Standard medical therapy: diuretics, lactulose, rifaximin, diuretics, albumin infusion, nutritional support (as required)
- Growth hormone + Standard medical therapy (Experimental): GH therapy will be initiated at a low dose of 2U/day and titrated slowly based on IGF-1 levels) subcutaneously for 1 year.
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — GH therapy will be initiated at a low dose of 2U/day and titrated slowly based on IGF-1 levels) subcutaneously for 1 year.
  Arms: Growth hormone + Standard medical therapy

SUMMARY:
Globally, cirrhosis and liver cancer carries a huge burden and accounts for about 3.5% (2 million) of all deaths every year. Once decompensated, i.e. development of ascites, variceal bleed, encephalopathy, and jaundice, the life expectancy is markedly reduced to a median of two years. The definitive treatment in this stage, i.e., liver transplantation is limited by cost, lack of donors, and life-long immunosuppression.

In addition to complications due to portal hypertension and hepatic insufficiency, decompensated cirrhosis is associated with malnutrition, sarcopenia, immune dysfunction, and impaired regeneration. Patients with cirrhosis are growth hormone (GH) resistant, with reduced insulin-like growth factor, which are linked to malnutrition and poor liver regeneration in cirrhosis. Diverse preclinical and clinical investigations in vitro and in vivo, have shown a benefit of GH in GH deficient, elderly and HIV positive patients. GH therapy in cirrhosis has been shown to improve nitrogen economy and to improve the GH resistance in a small pilot study by Donaghy et al. Also, GH therapy of short duration has shown to increase IGF1 levels, IGFBP-3 levels in patients of cirrhosis. GH therapy has also been shown to improve liver regeneration and protein synthesis after hepatectomy in patients of HCC with cirrhosis. However, there is a scarcity of data on clinical impact of long term administration of GH therapy in patients of cirrhosis. Hence, we undertook the present study to study the effect of growth hormone on clinical outcomes, malnutrition, immune cells and liver regeneration in patients with cirrhosis.

DETAILED DESCRIPTION:
Liver disease accounts for approximately 3.5% all deaths per year around the world, cirrhosis being the 11th most common cause of death globally. Liver cirrhosis is the final stage of all progressive and chronic liver diseases which progresses from asymptomatic compensated stage to decompensated at a rate of 5% to 7% each year. The major complications of liver cirrhosis are portal hypertension, ascites, spontaneous bacterial peritonitis (SBP), variceal bleed, hepatic encephalopathy (HE), hepatocellular carcinoma (HCC). Moreover, complications like protein-calorie malnutrition associated with sarcopenia, cirrhosis associated immune dysfunction (CAID) and impaired regeneration further adds to reduced survival. Liver transplantation is the only effective treatment for these patients but it is limited by resources, costs, expertise, and organ availability. Malnutrition is common in cirrhosis with prevalence ranging from 65 to 100%. Sarcopenia or loss of skeletal muscle mass is the major component of malnutrition in cirrhosis with prevalence of 40- 60%. Independent clinical consequences of sarcopenia in cirrhosis include lower survival, quality of life & increases risk of complications. Lack of improvement with nutritional supplementation is observed which may be attributed to GH resistance in cirrhotic patients further worsening sarcopenia.

CAID is a dynamic phenomenon, comprised of both increased systemic inflammation and immunodeficiency, ultimately leading to 30% mortality. Immunodeficiency in cirrhosis roots from deranged local immunity of liver, compromised immune surveillance of the liver and impairments in systemic immune cells (innate as well as adaptive).The systemic inflammation results from persistent immune cell stimulation due to enhanced gut translocation leading to increased production of various proinflammatory cytokines.

Liver regeneration is a complex and unique process. Hepatocytes have a remarkable capacity to meet the replacement demands during cellular loss. However, this regenerative capacity is overwhelmed during the late stage of acute liver injury, compromised in chronic liver injury, and lost in acute-on-chronic liver injury.

GH administration have been shown to improve sarcopenia, immune functions & regeneration in clinical studies and preclinical studies both in vitro and in vivo. Patients with chronic liver diseases are GH resistant i.e. they have high GH levels & low levels of IGF-1. So, in this study, we will investigate the impact of growth hormone on additional parameters including clinical outcomes, immunological profile and select parameters of liver regeneration in decompensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients having confirmed diagnosis of decompensated cirrhosis, any etiology.
3. Patients having given an informed and written consent for participation in the study.

Exclusion Criteria:

1. Acute on chronic liver failure.
2. Diagnosis of concomitant hepatocellular carcinoma or other active malignancy.
3. Severe cardiac dysfunction NYHA grade III/IV, Chronic obstructive pulmonary disease GOLD C or above.
4. Active alcohol abuse in last 3 months.
5. Known hypersensitivity to GH.
6. Human immunodeficiency virus seropositivity.
7. Patients on antiviral therapy for HCV, HBV or corticosteroid for autoimmune hepatitis those who have received it within the last 6 months.
8. TIPS insertion within 6 months prior to study inclusion.
9. Pregnancy & lactation.
10. Uncontrolled diabetes (Hb A1c ≥ 9) or diabetic retinopathy.
11. Active sepsis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Complication free survival | 12 Month
  Complications of cirrhosis - Ascites, Hepatic encephalopathy, Gastrointestinal bleeding, Bacterial infections, Acute kidney injury
Transplant free survival | 12 Month
  Transplant free survival where event is transplant or death
Incidence of complications of cirrhosis and infections | 12 Month
  Complications of cirrhosis - Ascites, Hepatic encephalopathy, Gastrointestinal bleeding, Bacterial infections, Acute kidney injury
Change in disease severity scores (CTP score) | 12 Month
  The Child-Turcotte-Pugh (CTP) score is used to assess the prognosis of patients with cirrhosis. The Pugh-Child score is determined by scoring five clinical measures of liver disease (Encephalopathy, Ascites, Albumin, Bilirubin and INR). A score of 1, 2, or 3 is given to each measure, with 3 being the most severe.
Change in disease severity scores (MELD Na) | 12 Month
  The MELD/Na score is a scoring system for accessing the severity of chronic liver disease using values as serum bilirubin, serum creatinine, and the international normalized ratio for prothrombin time and sodium, to predict survival.
Treatment related adverse events | 12 Month
  Any adverse events related to growth hormone

SECONDARY OUTCOMES:
Assessment of sarcopenia | 12 Month
  Sarcopenia will be assessed by calculation of Skeletal muscle index by taking cross sectional area of the psoas muscle at the level of the third lumbar vertebra on abdomen CT scans.
Change in liver frailty index | 12 Month
  LFI (Liver frailty index) will be calculated by FrAILT software©
Change in nitrogen balance | 12 Month
  Nitrogen balance will be calculated by using formula - Nitrogen intake - nitrogen output
Change in myostatin levels | 12 Month
  Myostatin in the serum will be measured in serum
Change in Functional capacity of Neutrophils | 12 Month
  Phagocytic capacity and oxidative burst of neutrophils will be assessed using flow cytometry
Immunophenotyping of neutrophils | 12 Month
  Immunophenotyping of neutrophils will be performed using flow-cytometry.
Change in cell death markers | 12 Month
  Markers of cell death - M30 & M65 will be assessed in serum using ELISA
Change in surrogate markers for hepatic regeneration | 12 Month
  surrogate markers for hepatic regeneration- Hepatocytes growth factor will be assessed in serum using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, DM, Study Director — Professor and Head, Department of Hepatology
Locations (1):
- Postgraduate Institute of Medical education and Research, Chandigarh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: No